CLINICAL TRIAL: NCT03577145
Title: Impact of Inulin on Production of Phenolic Acids From Tomato Onion and Lovage Soup
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Scottish Universities Environmental Research Centre (Other)
Responsible Party: Principal Investigator, Christine Edwards, Professor, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BB/MO27724/1-2
Record Dates: First submitted 2017-12-19; First posted 2018-07-05 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Healthy Adults
Keywords: Bioavailability; Polyphenols; Dietary fibre; Phenolic acids
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Intervention Model Description: Acute human bioavailability studies with a cross-over design. Subjects will be given a soup or drink in one of three combinations
  1. Tomato onion and lovage soup
  2. Inulin
  3. Mixture of tomato onion and lovage soup with inulin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tomato, onion & lovage soup with inulin (Experimental): One dose of tomato (300g), onion (100g) & lovage (20g) with 10g inulin will be given to subjects in the form of a soup
  Interventions: Dietary Supplement: Tomato, onion & lovage soup with inulin
- Tomato, onion & lovage soup (Experimental): One dose of tomato (300g), onion (100g) & lovage (20g) will be given to subjects in the form of a soup
  Interventions: Dietary Supplement: Tomato, onion & lovage soup
- Inulin (Experimental): One dose of 10g inulin will be given to subjects in the form of a drink
  Interventions: Dietary Supplement: Inulin

INTERVENTIONS:
Dietary Supplement: Tomato, onion & lovage soup with inulin — Source of polyphenols and non digestible carbohydrate
  Arms: Tomato, onion & lovage soup with inulin
Dietary Supplement: Tomato, onion & lovage soup — Source of polyphenols
  Arms: Tomato, onion & lovage soup
Dietary Supplement: Inulin — Source of non digestible carbohydrate
  Arms: Inulin

SUMMARY:
This is an acute human bioavailability study in self-reported healthy participants aged 20-70 years old. The investigators hypothesize that combination of polyphenolics from a soup rich in rutin and quercitin and the non-digestible carbohydrate (NDC) inulin will increase the production of phenolic acids by bacteria in the human colon and these will be detected in urine. Participants will attend for three arms in a randomized order: Tomato, onion and lovage soup (high polyphenol food), Inulin (NDC) or Mixture of tomato, onion and lovage soup and inulin.

During each feeding study, urine, blood and stool samples will be collected at regular intervals for the duration of 24 hrs after consumption of test food. Participants will be asked to follow a low polyphenol diet for 2 days prior to the feeding study.

DETAILED DESCRIPTION:
Polyphenol rich plant foods have been associated with several health benefits but their bioavailability is generally low. The majority of plant polyphenols are poorly absorbed in the small intestine and enter the colon where the colonic microbiota metabolise them to release a range of phenolic acids, which are now thought to be the main bioactive components related to the reduction in disease risk. Very little is known about the impact of other constituents of the diet on the metabolism and bacterial catabolism of these polyphenols.

Colonic bacteria are key agents in the release of the bioactive molecules from polyphenols but also ferment non-digestible carbohydrates (NDC) such as inulin to short chain fatty acids. It is likely that there are key interactions in the colonic bacterial metabolism of NDC and phenolics. The investigators hypothesize that combination of polyphenolics (in onions, tomatoes and lovage) with inulin (NDC) will increase the urinary output of bioactive phenolic acids.

ELIGIBILITY:
Inclusion Criteria:

• Self-reported healthy adults

Exclusion Criteria:

* Antibiotic use within the last 3 months
* Identified gastro-intestinal diseases
* On prescribed medication other than the contraceptive pill
* Pregnant or breastfeeding.
* Diagnosed as anaemic
* Allergic to paracetamol or any food

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Phenolic acids bioavailability | 0-24 hrs
  Urine excretion of phenolic acids (µg) will be measured with GC-MS

SECONDARY OUTCOMES:
Glycaemic measurements | 0-8 hrs
  Plasma glucose (mmol/L), insulin (mU/L) will be measured by commercial kits
Appetite hormones measurements | 0-8 hrs
  Appetite hormone (PYY) levels in plasma (pg/mL) will be measured by commercial Elisa kit
Mouth to caecum transit time | 0-8 hrs
  Mouth to caecum transit time (in hours/mins) will be calculated from sustained rise in breath hydrogen level measurements by hydrogen monitor
Gastric emptying time | 0-6 hrs
  Gastric emptying time (in hours/mins) will be estimated using kinetics of plasma paracetamol levels measured by acetaminophen assay kits

CONTACTS AND LOCATIONS:
Overall Officials: Christine Edwards, PhD, Principal Investigator — University of Glasgow
Locations (1):
- School of Medicine, Nursing and Dentistry, College of MVLS, University of Glasgow, Glasgow, Lanarkshire, United Kingdom

REFERENCES:
- [Background] Russell W, Duthie G. Plant secondary metabolites and gut health: the case for phenolic acids. Proc Nutr Soc. 2011 Aug;70(3):389-96. doi: 10.1017/S0029665111000152. PMID 21781364
- [Background] Roowi S, Mullen W, Edwards CA, Crozier A. Yoghurt impacts on the excretion of phenolic acids derived from colonic breakdown of orange juice flavanones in humans. Mol Nutr Food Res. 2009 May;53 Suppl 1:S68-75. doi: 10.1002/mnfr.200800287. PMID 19415668
- [Background] Tamura M, Nakagawa H, Tsushida T, Hirayama K, Itoh K. Effect of pectin enhancement on plasma quercetin and fecal flora in rutin-supplemented mice. J Food Sci. 2007 Nov;72(9):S648-51. doi: 10.1111/j.1750-3841.2007.00557.x. PMID 18034749

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT03577145/Prot_SAP_000.pdf